CLINICAL TRIAL: NCT00023673
Title: A Phase I/II Dose Intensification Study Using Three Dimensional Conformal Radiation Therapy And Concurrent Chemotherapy For Patients With Inoperable, Non-Small Cell Lung Cancer
Brief Title: Radiation Therapy Combined With Paclitaxel and Carboplatin in Treating Patients With Stage III Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTOG L-0117; CDR0000068850 (Registry Identifier: PDQ (Physician Data Query)); NCI-2012-02401 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2001-09-13; First posted 2003-04-09 (Estimated); Results first posted 2014-03-27 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-11

CONDITIONS: Lung Cancer
Keywords: squamous cell lung cancer; large cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; adenocarcinoma of the lung; adenosquamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Carboplatin; Paclitaxel

ARMS (4):
- Phase I: 75.25 Gy/36 fx + chemotherapy (Experimental): Phase I: Three-dimensional conformal radiation therapy (3DRT) of 75.25 Gy given in 36 fractions (2.15 Gy per fraction) with concurrent chemotherapy consisting of weekly paclitaxel at 50mg/m2 and carboplatin at area under the curve 2mg/m2. Adjuvant systemic chemotherapy (two cycles of paclitaxel and carboplatin) following completion of RT was optional.
  Interventions: Drug: carboplatin; Drug: paclitaxel; Radiation: three-dimensional conformal radiation therapy
- Phase I: 74 Gy/37 fx + chemotherapy (Experimental): Phase I: Three-dimensional conformal radiation therapy (3DRT) of 74 Gy given in 37 fractions (2.0 Gy per fraction) with concurrent chemotherapy consisting of weekly paclitaxel at 50mg/m2 and carboplatin at area under the curve 2mg/m2. Adjuvant systemic chemotherapy (two cycles of paclitaxel and carboplatin) following completion of RT was optional.
  Interventions: Drug: carboplatin; Drug: paclitaxel; Radiation: three-dimensional conformal radiation therapy
- Phase I: 70 Gy/35 fx + chemotherapy (Experimental): Phase I: Three-dimensional conformal radiation therapy (3DRT) of 70 Gy given in 35 fractions (2.0 Gy per fraction) with concurrent chemotherapy consisting of weekly paclitaxel at 50mg/m2 and carboplatin at area under the curve 2mg/m2. Adjuvant systemic chemotherapy (two cycles of paclitaxel and carboplatin) following completion of RT was optional.
  Interventions: Drug: carboplatin; Drug: paclitaxel; Radiation: three-dimensional conformal radiation therapy
- Phase II: 74 Gy/37 fx + chemotherapy (Experimental): Phase II: Three-dimensional conformal radiation therapy (3DRT) of 74 Gy given in 37 fractions (2.0 Gy per fraction) with concurrent chemotherapy consisting of weekly paclitaxel at 50mg/m2 and carboplatin at area under the curve 2mg/m2. Adjuvant systemic chemotherapy (two cycles of paclitaxel and carboplatin) following completion of RT was optional.
  Interventions: Drug: carboplatin; Drug: paclitaxel; Radiation: three-dimensional conformal radiation therapy

INTERVENTIONS:
Drug: carboplatin
Drug: paclitaxel
Radiation: three-dimensional conformal radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and giving them with specialized radiation therapy may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the effectiveness of radiation therapy combined with paclitaxel and carboplatin in treating patients who have stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of 3-dimensional conformal radiotherapy when administered concurrently with paclitaxel and carboplatin in patients with inoperable stage IIIA or IIIB non-small cell lung cancer. (Phase I) (Closed to accrual as of 01/13/04.)
* Determine the 12-month survival rate in patients treated with this regimen. (Phase II) (Closed to accrual as of 11/27/07.)
* Determine the toxicity of this regimen in these patients.
* Determine the partial organ tolerance doses for the lung and esophagus in patients treated with this regimen.
* Determine the complete response rate in patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of 3-dimensional conformal radiotherapy.

* Phase I (closed to accrual as of 01/13/04): Patients undergo 3-dimensional conformal radiotherapy once daily five days a week for 7-8 weeks. Patients also receive concurrent chemotherapy comprising paclitaxel IV over 1 hour followed by carboplatin IV over 30 minutes on days 1, 8, 15, 22, 29, 36, and 43.

Cohorts of 7-9 patients receive de-escalating doses of 3-dimensional conformal radiotherapy until the maximum tolerated dose (MTD) is determined when given in combination with chemotherapy. The MTD is defined as the highest dose at which no more than 1 patient experiences dose-limiting toxicity.

* Phase II: Additional patients are accrued and treated as above at the MTD. At least 3 weeks after completing radiotherapy, patients may receive additional chemotherapy comprising paclitaxel IV over 3 hours once and carboplatin IV over 30 minutes once. Treatment with paclitaxel and carboplatin may repeat every 3 weeks for up to 2 courses.

Patients are followed every 3 months for 1 year, every 4 months for 1 year, every 6 months for 3-5 years, and then annually thereafter.

PROJECTED ACCRUAL: A maximum of 73 patients (up to 27 for phase I [closed to accrual as of 10/28/04] and 46 for phase II) will be accrued for this study within 1-1.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed unresectable stage IIIB non-small cell lung cancer

  * Squamous cell carcinoma
  * Adenocarcinoma
  * Large cell carcinoma
  * Non-small cell carcinoma not otherwise specified
* All detectable primary tumor and involved regional lymph nodes must be encompassed by radiotherapy fields
* Measurable disease on 3-dimensional planning CT scan
* No undifferentiated small cell (oat cell or high-grade neuroendocrine) carcinoma
* No stage IV or recurrent disease
* No distant metastases or supraclavicular lymph node involvement
* No significant atelectasis (i.e., atelectasis of an entire lung)
* No pleural effusions, pericardial effusions, or superior vena cava syndrome
* No lung cancer within the past 2 years
* Ineligible for currently open Radiation Therapy Oncology Group (RTOG) phase III lung protocols

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Zubrod 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin less than 1.5 mg/dL
* Aspartate aminotransferase (AST) less than 2 times upper limit of normal

Renal:

* Creatinine no greater than 2.0 mg/dL

Pulmonary:

* Forced expiratory volume (FEV)_1 at least 1.0 L

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No weight loss greater than 5% in the past 6 months
* No other malignancy within the past year except nonmelanoma skin cancer
* Completed 3D plan with total lung V20 </= 30% mean esophageal dose </= 34 Gy and esophageal V55 </= 30%

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior biologic response modifiers for current lung cancer
* At least 5 years since prior biologic response modifiers

Chemotherapy:

* No prior chemotherapy for current lung cancer
* At least 5 years since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy to the thorax

Surgery:

* No prior complete tumor resection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2001-07; Primary Completion 2009-01 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Bradley, MD, Study Chair — Mallinckrodt Institute of Radiology at Washington University Medical Center
Locations (41):
- United States (40):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Arizona Oncology Services Foundation, Phoenix, Arizona
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Providence Holy Cross Cancer Center, Mission Hills, California
  - University of California Davis Cancer Center, Sacramento, California
  - Bay Medical, Panama City, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Alexian Brothers Radiation Oncology, Elk Grove Village, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Oncology Center at Saint Margaret Mercy Healthcare Center, Hammond, Indiana
  - Cancer Center at Ball Memorial Hospital, Muncie, Indiana
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Cancer Institute of Cape Girardeau, LLC, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - Ocean Medical Center at Meridian Health, Brick, New Jersey
  - J. Phillip Citta Regional Cancer Center at Community Medical Center, Toms River, New Jersey
  - Franklin & Edith Scarpa Regional Cancer Center at South Jersey Healthcare, Vineland, New Jersey
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - High Point Regional Hospital, High Point, North Carolina
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Three Rivers Community Hospital, Grants Pass, Oregon
  - Dubs Cancer Center at Rogue Valley Medical Center, Medford, Oregon
  - Providence Cancer Center at PMCC, Medford, Oregon
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - University of Texas Medical Branch, Galveston, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Schiffler Cancer Center at Wheeling Hospital, Wheeling, West Virginia
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee, Milwaukee, Wisconsin
- Tom Baker Cancer Centre - Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Result] Bradley JD, Bae K, Graham MV, Byhardt R, Govindan R, Fowler J, Purdy JA, Michalski JM, Gore E, Choy H. Primary analysis of the phase II component of a phase I/II dose intensification study using three-dimensional conformal radiation therapy and concurrent chemotherapy for patients with inoperable non-small-cell lung cancer: RTOG 0117. J Clin Oncol. 2010 May 10;28(14):2475-80. doi: 10.1200/JCO.2009.27.1205. Epub 2010 Apr 5. PMID 20368547
- [Result] Bradley JD, Moughan J, Graham MV, Byhardt R, Govindan R, Fowler J, Purdy JA, Michalski JM, Gore E, Choy H. A phase I/II radiation dose escalation study with concurrent chemotherapy for patients with inoperable stages I to III non-small-cell lung cancer: phase I results of RTOG 0117. Int J Radiat Oncol Biol Phys. 2010 Jun 1;77(2):367-72. doi: 10.1016/j.ijrobp.2009.04.029. PMID 20457350
- [Result] Bradley JD, Graham M, Suzanne S, et al.: Phase I results of RTOG L-0117: a phase I/II dose intensification study using 3DCRT and concurrent chemotherapy for patients with inoperable NSCLC. [Abstract] J Clin Oncol 23 (Suppl 16): A-7063, 636s, 2005.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phase I: 75.25 Gy/36 fx + Chemotherapy | Phase I: 74 Gy/37 fx + Chemotherapy | Phase I: 70 Gy/35 fx + Chemotherapy | Phase II: 74 Gy/37 fx + Chemotherapy
Started | 8 | 9 | 0 | 46
Completed | 8 (Phase I eligible patients starting protocol treatment are considered to have completed the study.) | 9 (Phase I eligible patients starting protocol treatment are considered to have completed the study.) | 0 (This arm was not used since further de-escalation was not required.) | 44 (Phase II subjects contributing data to primary analysis are considered to have completed the study.)
Not Completed | 0 | 0 | 0 | 2
Not completed — Ineligible / no protocol treatment | 0 | 0 | 0 | 1
Not completed — Patient withdrew consent | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Eligible patients who started protocol treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: 75.25 Gy/36 fx + Chemotherapy | Phase I: 74 Gy/37 fx + Chemotherapy | Phase II: 74 Gy/37 fx + Chemotherapy | Total
Number analyzed (Participants) | 8 | 9 | 44 | 61
Age, Continuous [Median (Full Range); unit: years] | 65.5 [48 to 77] | 68 [52 to 81] | 67 [43 to 83] | 67 [43 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 8 | 7 | 16
  Male | 7 | 1 | 37 | 45

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Three-dimensional Conformal Radiation Therapy (3DRT), in Terms of Gy Per Fraction, Combined With Concurrent Chemotherapy
Description: Dose limiting toxicity (DLT) = Grade 3/4 non-hematologic toxicities (excluding nausea, vomiting, and alopecia) and Grade 4 hematologic toxicities. The DLT rate for this study was set at 40% based on Radiation Therapy Oncology Group (RTOG) study 94-10. No acute (within 90 days from start of 3DRT) DLT's in the first 5 patients (0/5) or the combination of one acute DLT in the first 5 patients (1/5) and none in the next 2 patients (0/2) was required to deem a given dose level to be acceptable. If at any time a Grade 5 toxicity (death) occurred, accrual would be suspended and the event reviewed by a study chair. At any given dose level, this design gives at least 90% confidence that the true acute DLT rate is less than 40% and the probability of not escalating when the true toxicity rate is 40% or higher is at least 83%.
  Rating scale: 0 = not the MTD, 1 = MTD
Time Frame: From start of treatment to 90 days
Population: The first seven eligible patients who started protocol treatment at each dose level.
Measure: Number; unit: units on a scale
Arm/Group | Phase I: 75.25 Gy/36 fx + Chemotherapy | Phase I: 74 Gy/37 fx + Chemotherapy
Number analyzed (Participants) | 7 | 7
units on a scale | 0 | 1

2. Primary Outcome: Percentage of Patients Who Survive at Least 12 Months
Description: Null hypothesis: p<= 62.3% (the best arm of RTOG 94-10); alternative hypothesis: p>= 77.9%. Where p is the percentage of patients alive at at 12 months. Using a one-group chi-square test with alpha = 0.10, a sample size of 50 patients provides at least 87% power to detect a 25% or greater relative increase in the 12-month survival rate, or equivalently, an absolute increase of at least 15.6 percentage points (62.3 versus 77.9). If the point estimate is greater than 71.1% (upper bound), then the conclusion is that the 12-month survival rate from the new treatment significantly improved from 62.3%.
Time Frame: From registration to 1 year
Population: Eligible patients at the MTD dose level who started protocol treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase I/II: 74 Gy/37 fx + Chemotherapy: Phase I/II: Three-dimensional conformal radiation therapy (3DRT) of 74 Gy given in 37 fractions (2.0 Gy per fraction) with concurrent chemotherapy consisting of weekly paclitaxel at 50mg/m2 and carboplatin at area under the curve 2mg/m2. Adjuvant systemic chemotherapy (two cycles of paclitaxel and carboplatin) following completion of RT was optional.
  carboplatin
  paclitaxel
  three-dimensional conformal radiation therapy
Arm/Group | Phase I/II: 74 Gy/37 fx + Chemotherapy
Number analyzed (Participants) | 53
percentage of participants | 75.5 [61.5 to 85.0]

3. Secondary Outcome: Frequency of Highest Grade Chemotherapy/Acute RT Toxicities and Late RT Toxicities.
Description: Highest grade toxicity per subject was counted. Toxicities were graded using the Common Toxicity Criteria (CTC) v 2.0 for chemotherapy/acute RT toxicities and using the RTOG/EORTC Late Toxicity Criteria for late RT toxicity. Grade refers to the severity of the toxicity. Both criteria assign Grades 1 through 5 with unique clinical descriptions of severity for a given toxicity based on this general guideline: Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening or disabling, Grade 5 Death related to toxicity.Chemotherapy/Acute RT toxicities occur during chemotherapy and/or within 90 days of the start of RT. Late RT toxicities occur more than 90 days after the start of RT.
Time Frame: Chemotherapy/Acute RT toxicity: from start of treatment to 90 days from start of study treatment; Late RT toxicity: from 90 days after start of treatment to last follow-up (Maximum follow-up = 57.9 months.)
Population: Eligible patients from Phase I and II 74 Gy arms who started study treatment. Additionally for late RT toxicity, those who have toxicity data at least 90 days from start of RT.
Measure: Count of Participants; unit: Participants
Groups:
- Phase I/II: 74 Gy/37 fx + Chemotherapy: Phase I/II: Three-dimensional conformal radiation therapy (3DRT) of 74 Gy given in 37 fractions (2.0 Gy per fraction) with concurrent chemotherapy consisting of weekly paclitaxel at 50mg/m2 and carboplatin at area under the curve 2mg/m2. Adjuvant systemic chemotherapy (two cycles of paclitaxel and carboplatin) following completion of RT was optional.
Arm/Group | Phase I/II: 74 Gy/37 fx + Chemotherapy
Number analyzed (Participants) | 53
Participants
  Chemotherapy/Acute RT non-hematologic: Grade 1 | 4
  Chemotherapy/Acute RT non-hematologic: Grade 2 | 16
  Chemotherapy/Acute RT non-hematologic: Grade 3 | 28
  Chemotherapy/Acute RT non-hematologic: Grade 4 | 2
  Chemotherapy/Acute RT non-hematologic: Grade 5 | 2
  Chemotherapy/Acute RT hematologic: Grade 1 | 1
  Chemotherapy/Acute RT hematologic: Grade 2 | 8
  Chemotherapy/Acute RT hematologic: Grade 3 | 37
  Chemotherapy/Acute RT hematologic: Grade 4 | 5
  Chemotherapy/Acute RT hematologic: Grade 5 | 2
  Late RT toxicity: Grade 1: number analyzed (Participants) | 50
  Late RT toxicity: Grade 1 | 13
  Late RT toxicity: Grade 2: number analyzed (Participants) | 50
  Late RT toxicity: Grade 2 | 10
  Late RT toxicity: Grade 3: number analyzed (Participants) | 50
  Late RT toxicity: Grade 3 | 9
  Late RT toxicity: Grade 4: number analyzed (Participants) | 50
  Late RT toxicity: Grade 4 | 1
  Late RT toxicity: Grade 5: number analyzed (Participants) | 50
  Late RT toxicity: Grade 5 | 1

4. Secondary Outcome: Partial Organ Tolerance Doses for Lung and Esophagus (Percent Volume of Total Lung Receiving > 20 Gy by Toxicity Level)
Description: Percent volume of total lung receiving > 20 Gy radiation therapy (Lung V20) was compared between the two patient groups of those who experienced a grade 3 and higher lung toxicity and those who did not. Similarly, it was also compared between the two patient groups of those who experienced a grade 2 and higher esophageal toxicity and those who did not. Toxicities graded using CTC v 2.0 for chemotherapy/acute RT toxicities and using the RTOG/EORTC Late Toxicity Criteria for late RT toxicity. Grade refers to the severity of the toxicity. Both criteria assign Grades 1 through 5 with unique clinical descriptions of severity for a given toxicity based on this general guideline: Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening or disabling, Grade 5 Death related to toxicity.
Time Frame: From start of treatment to last follow-up (Maximum follow-up = 57.9 months.)
Population: All eligible patients on the phase I and II 74 Gy arms who received treatment and had RT plan data available with the given structure
Measure: Median (Full Range); unit: Percent (V20)
Groups:
- No High Grade Toxicity: For lung toxicity, no high grade toxicity means < Grade 3. For esophagitis toxicity, no high grade toxicity means < Grade 2. Therefore overall number of participants analyzed differs.
- High Grade Toxicity: For lung toxicity, high grade toxicity means >= Grade 3. For esophagitis toxicity, high grade toxicity means >= Grade 2. Therefore overall number of participants analyzed differs.
Arm/Group | No High Grade Toxicity | High Grade Toxicity
Number analyzed (Participants) | 53 | 53
Percent (V20)
  Lung Toxicity: Lung V20: number analyzed (Participants) | 39 | 12
  Lung Toxicity: Lung V20 | 24.1 [9.9 to 35.7] | 26.3 [15.6 to 33.3]
  Esophagitis Toxicity: Lung V20: number analyzed (Participants) | 30 | 21
  Esophagitis Toxicity: Lung V20 | 22.4 [9.9 to 35.7] | 26.3 [14.0 to 33.3]
Statistical Analysis 1: Comparison: No High Grade Toxicity vs High Grade Toxicity; Lung toxicity (<Grade 3 vs. >= Grade 3): Lung V20; Test type: Superiority; p = 0.62, Wilcoxon (Mann-Whitney); 2-sided significance level = 0.05
Statistical Analysis 2: Comparison: No High Grade Toxicity vs High Grade Toxicity; Esophagitis toxicity (<Grade 2 vs. >= Grade 2): Lung V20; Test type: Superiority; p = 0.22, Wilcoxon (Mann-Whitney); 2-sided significance level = 0.05

5. Secondary Outcome: Partial Organ Tolerance Doses for Lung and Esophagus (Mean Organ Dose by Toxicity Level)
Description: Mean lung dose was compared between the two patient groups of those who experienced a grade 3 and higher lung toxicity and those who did not. Similarly, mean lung dose, and mean esophageal dose were compared between the two patient groups of those who experienced a grade 2 and higher esophageal toxicity and those who did not. Toxicities graded using CTC v 2.0 for chemotherapy/acute RT toxicities and using the RTOG/EORTC Late Toxicity Criteria for late RT toxicity. Grade refers to the severity of the toxicity. Both criteria assign Grades 1 through 5 with unique clinical descriptions of severity for a given toxicity based on this general guideline: Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening or disabling, Grade 5 Death related to toxicity.
Time Frame: From start of treatment to last follow-up (Maximum follow-up = 57.9 months.)
Population: as for outcome 4
Measure: Mean (Full Range); unit: Gy (mean dose)
Arm/Group | No High Grade Toxicity | High Grade Toxicity
Number analyzed (Participants) | 53 | 53
Gy (mean dose)
  Lung Toxicity: Mean Lung Dose: number analyzed (Participants) | 39 | 12
  Lung Toxicity: Mean Lung Dose | 15.2 [5.7 to 21.8] | 17.2 [11.5 to 18.9]
  Esophagitis Toxicity: Mean Lung Dose: number analyzed (Participants) | 30 | 21
  Esophagitis Toxicity: Mean Lung Dose | 14.5 [5.7 to 21.8] | 16.9 [9.9 to 20.6]
  Esophagitis Toxicity: Mean Esophageal Dose: number analyzed (Participants) | 30 | 22
  Esophagitis Toxicity: Mean Esophageal Dose | 21.0 [7.1 to 34.9] | 24.6 [16.2 to 33.7]
Statistical Analysis 1: Comparison: No High Grade Toxicity vs High Grade Toxicity; Lung toxicity (<Grade 3 vs. >= Grade 3): Mean Lung Dose; Test type: Superiority; p = 0.30, t-test, 2 sided; 2-sided significance level = 0.05
Statistical Analysis 2: Comparison: No High Grade Toxicity vs High Grade Toxicity; Esophagitis toxicity (<Grade 2 vs. >= Grade 2): Mean Lung Dose; Test type: Superiority; p = 0.17, t-test, 2 sided; 2-sided significance level = 0.05
Statistical Analysis 3: Comparison: No High Grade Toxicity vs High Grade Toxicity; Esophagitis toxicity (<Grade 2 vs. >= Grade 2): Mean Esophageal Dose; Test type: Superiority; p = 0.08, t-test, 2 sided; 2-sided significance level = 0.05

6. Secondary Outcome: Number of Patients With Complete Response at 3 Months After Completion of Therapy
Description: "Complete response" means no evidence of tumor on the CT scan.
Time Frame: From start of treatment until 3 months after completion of all study treatment, estimated to be 5 or 6.5 months depending whether or not subject received optional adjuvant chemotherapy.
Population: Eligible patients from Phase I and II 74 Gy arms who started study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I/II: 74 Gy/37 fx + Chemotherapy
Number analyzed (Participants) | 53
Participants | 3

ADVERSE EVENTS:
Description: Subjects experiencing more than one of a given serious adverse event (SAE) are counted only once for that SAE. The same methodology was applied for non-SAE adverse events (AE).
Groups:
- Phase I/II: 74 Gy/37 fx + Chemotherapy: Phase I: Three-dimensional conformal radiation therapy (3DRT) of 74 Gy given in 37 fractions (2.0 Gy per fraction) with concurrent chemotherapy consisting of weekly paclitaxel at 50mg/m2 and carboplatin at area under the curve 2mg/m2. Adjuvant systemic chemotherapy (two cycles of paclitaxel and carboplatin) following completion of RT was optional.
Arm/Group | Phase I: 75.25 Gy/36 fx + Chemotherapy | Phase I/II: 74 Gy/37 fx + Chemotherapy
Serious Adverse Events (participants affected / at risk) | 7/8 | 36/53
Other Adverse Events (participants affected / at risk) | 8/8 | 52/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: 75.25 Gy/36 fx + Chemotherapy (N=8) | Phase I/II: 74 Gy/37 fx + Chemotherapy (N=53)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 | 1
Hemolysis NOS (Blood and lymphatic system disorders) | 0 | 1
Packed red blood cell transfusion (Blood and lymphatic system disorders) | 0 | 1
Platelet transfusion (Blood and lymphatic system disorders) | 0 | 1
Arrhythmia NOS (Cardiac disorders) | 0 | 2
Sinus tachycardia (Cardiac disorders) | 1 | 0
Supraventricular arrhythmia NOS (Cardiac disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Esophageal spasm (Gastrointestinal disorders) | 0 | 3
Esophagitis NOS (Gastrointestinal disorders) | 0 | 2
GI-other (Gastrointestinal disorders) | 0 | 2
Ileus (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Vomiting NOS (Gastrointestinal disorders) | 0 | 2
Late RT Toxicity: Esophagus (General disorders) | 0 | 4
Late RT Toxicity: Heart (General disorders) | 0 | 1
Late RT Toxicity: Lung (General disorders) | 1 | 8
Late RT Toxicity: Other (General disorders) | 1 | 0
Pain-other (General disorders) | 1 | 0
Hypersensitivity NOS (Immune system disorders) | 1 | 2
Infection NOS (Infections and infestations) | 1 | 5
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 0 | 1
Infection with unknown ANC (Infections and infestations) | 0 | 1
Infection, Other (Infections and infestations) | 0 | 1
Dermatitis radiation NOS (Injury, poisoning and procedural complications) | 0 | 1
Operative injury of vein/artery (Injury, poisoning and procedural complications) | 0 | 1
Cardiac troponin I increased (Investigations) | 1 | 0
Leukopenia NOS (Investigations) | 1 | 19
Lymphopenia (Investigations) | 0 | 1
Neutropenia (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Hyperglycemia NOS (Metabolism and nutrition disorders) | 1 | 4
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 1 | 0
Convulsions NOS (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 2
Renal failure NOS (Renal and urinary disorders) | 0 | 1
Renal/GU-Other (Renal and urinary disorders) | 0 | 1
Dyspnea NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary-other (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypotension NOS (Vascular disorders) | 0 | 2
Peripheral ischaemia NOS (Vascular disorders) | 0 | 1
Thrombosis NOS (Vascular disorders) | 0 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: 75.25 Gy/36 fx + Chemotherapy (N=8) | Phase I/II: 74 Gy/37 fx + Chemotherapy (N=53)
Hematologic-Other (Blood and lymphatic system disorders) | 0 | 6
Hemoglobin decreased (Blood and lymphatic system disorders) | 5 | 34
Pericardial effusion (Cardiac disorders) | 0 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 3
Supraventricular arrhythmia NOS (Cardiac disorders) | 0 | 3
Hearing-Other (Ear and labyrinth disorders) | 0 | 3
Abdominal pain NOS (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 22
Diarrhea NOS (Gastrointestinal disorders) | 1 | 9
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 9
Dysphagia (Gastrointestinal disorders) | 1 | 3
Esophageal spasm (Gastrointestinal disorders) | 3 | 17
Esophagitis NOS (Gastrointestinal disorders) | 2 | 19
GI-other (Gastrointestinal disorders) | 1 | 2
Gastritis NOS (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 17
Radiation mucositis (Gastrointestinal disorders) | 0 | 4
Rectal bleeding (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 4
Vomiting NOS (Gastrointestinal disorders) | 1 | 9
Chest pain (General disorders) | 0 | 3
Edema NOS (General disorders) | 1 | 2
Fatigue (General disorders) | 2 | 40
Late RT Toxicity: Bone (General disorders) | 1 | 1
Late RT Toxicity: Esophagus (General disorders) | 4 | 9
Late RT Toxicity: Heart (General disorders) | 1 | 4
Late RT Toxicity: Lung (General disorders) | 5 | 26
Late RT Toxicity: Other (General disorders) | 2 | 8
Late RT Toxicity: Skin (within the irradiated field) (General disorders) | 1 | 5
Late RT Toxicity: Spinal cord (General disorders) | 1 | 1
Late RT Toxicity: Subcutaneous tissue (General disorders) | 1 | 2
Pain due to radiation (General disorders) | 0 | 11
Pain-other (General disorders) | 1 | 13
Pyrexia (General disorders) | 0 | 9
Rigors (General disorders) | 0 | 1
Hepatic-Other (Hepatobiliary disorders) | 0 | 4
Hypersensitivity NOS (Immune system disorders) | 0 | 1
Infection NOS (Infections and infestations) | 2 | 2
Infection with unknown ANC (Infections and infestations) | 0 | 1
Dermatitis radiation NOS (Injury, poisoning and procedural complications) | 2 | 14
Activated partial thromboplastin time prolonged (Investigations) | 0 | 2
Alanine aminotransferase increased (Investigations) | 1 | 6
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood alkaline phosphatase NOS increased (Investigations) | 2 | 3
Blood bilirubin increased (Investigations) | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 5
Forced expiratory volume decreased (Investigations) | 0 | 1
Leukopenia NOS (Investigations) | 6 | 29
Lymphopenia (Investigations) | 2 | 17
Metabolic-Other (Investigations) | 0 | 2
Neutropenia (Investigations) | 2 | 25
Platelet count decreased (Investigations) | 2 | 20
Prothrombin time prolonged (Investigations) | 1 | 3
Weight decreased (Investigations) | 2 | 13
Anorexia (Metabolism and nutrition disorders) | 2 | 21
Blood albumin decreased (Metabolism and nutrition disorders) | 1 | 8
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 0 | 1
Blood magnesium decreased (Metabolism and nutrition disorders) | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 5
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia NOS (Metabolism and nutrition disorders) | 3 | 6
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 2
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 4
Hypoglycaemia NOS (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Joint, muscle, or bone-Other (Musculoskeletal and connective tissue disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 4
Amnesia NEC (Nervous system disorders) | 0 | 1
Ataxia NEC (Nervous system disorders) | 0 | 1
Convulsions NOS (Nervous system disorders) | 2 | 0
Dizziness (exc vertigo) (Nervous system disorders) | 1 | 5
Headache NOS (Nervous system disorders) | 1 | 4
Neuralgia NOS (Nervous system disorders) | 0 | 2
Neurologic-Other (Nervous system disorders) | 0 | 3
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 8
Speech disorder NEC (Nervous system disorders) | 0 | 1
Taste disturbance (Nervous system disorders) | 0 | 5
Tremor NEC (Nervous system disorders) | 0 | 1
Anxiety NEC (Psychiatric disorders) | 0 | 5
Confusion (Psychiatric disorders) | 0 | 2
Depression NEC (Psychiatric disorders) | 0 | 5
Insomnia NEC (Psychiatric disorders) | 0 | 12
Libido decreased (Psychiatric disorders) | 0 | 1
Renal failure NOS (Renal and urinary disorders) | 0 | 1
Renal/GU-Other (Renal and urinary disorders) | 0 | 2
Ureteric obstruction (Renal and urinary disorders) | 0 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 24
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Dyspnea NOS (Respiratory, thoracic and mediastinal disorders) | 2 | 18
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumothorax NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary-other (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 10
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 2 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Nail abnormality NOS (Skin and subcutaneous tissue disorders) | 0 | 3
Skin discoloration (Skin and subcutaneous tissue disorders) | 0 | 1
Skin-Other (Skin and subcutaneous tissue disorders) | 1 | 1
Flushing (Vascular disorders) | 0 | 1
Hypertension NOS (Vascular disorders) | 0 | 1
Hypotension NOS (Vascular disorders) | 0 | 3

LIMITATIONS AND CAVEATS:
This study was originally designed to escalate 3DRT via increasing doses per fraction. However, due to excessive toxicity at dose level 1 (75.25 Gy, 2.15 Gy/fraction), the protocol was amended in January 2003 to de-escalate 3DRT dose.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No